CLINICAL TRIAL: NCT01449188
Title: A Randomized, Double-blind, Four-period Crossover Study to Investigate the Effect of Intravenous Ondansetron, a 5-HT3 Antagonist, on Cardiac Conduction as Compared to Placebo and Moxifloxacin in Healthy Adult Subjects
Brief Title: To Investigate the Effect of Intravenous Ondansetron on Cardiac Conduction as Compared to Placebo and Moxifloxacin in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 115458
Record Dates: First submitted 2011-09-29; First posted 2011-10-10 (Estimated); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Nausea and Vomiting, Chemotherapy-Induced
Keywords: ondansetron; moxifloxacin; Zofran; thorough QT study; IV
MeSH Terms: conditions — Nausea; Vomiting | interventions — Ondansetron; Moxifloxacin; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- ondansetron, 8 mg IV over 15 minutes (Active Comparator): the lower ondansetron IV dose will be used in one of the four treatment periods
  Interventions: Drug: ondansetron
- ondansetron, 32 mg IV over 15 minutes (Active Comparator): the higher ondansetron IV dose will be used in one of the four treatment periods
  Interventions: Drug: ondansetron
- placebo for ondansetron, IV over 15 minutes (Placebo Comparator): placebo for ondansetron IV dose will be used in one of the four treatment periods
  Interventions: Other: saline
- moxifloxacin, 400mg tablet (oral) (Active Comparator): moxifloxacin is known to produce mild QT prolongation and will be used in one of the four treatment periods
  Interventions: Drug: moxifloxacin

INTERVENTIONS:
Drug: ondansetron — FDA approved drug used to treat nausea and vomiting
  Other Names: Zofran
  Arms: ondansetron, 32 mg IV over 15 minutes; ondansetron, 8 mg IV over 15 minutes
Drug: moxifloxacin — FDA approved antibiotic commonly used as a positive control in thorough QT studies
  Other Names: Avelox
  Arms: moxifloxacin, 400mg tablet (oral)
Other: saline — USP saline IV solution used as placebo for ondansetron IV.
  Arms: placebo for ondansetron, IV over 15 minutes

SUMMARY:
Ondansetron, also known as Zofran, is a marketed compound used for the prevention of nausea and vomiting. This study, called a thorough QT study, will characterize the effects of a single intravenous (IV) dose of ondansetron on cardiac repolarization as compared to placebo. Moxifloxacin, a commercially available antibiotic known to cause a mild QT prolongation, will be used as a positive control and will be given orally. The cardiac repolarization will be measured by taking consecutive ECGs on a recording device known as a Holter monitor and measuring the QT interval at specified times. In addition, blood samples will also be taken at specified times and will be used to measure the amount of study medication in the body.

DETAILED DESCRIPTION:
Ondansetron was first approved in 1991 for treatment of nausea and vomiting associated with chemotherapy and surgical procedures and as ondansetron was developed prior to current regulatory requirements, a formal, thorough QT study has not been performed for this compound. The purpose of this study is to further define the safety of ondansetron as some effects on QT interval prolongation have been observed for this and other members of the 5-HT3 inhibitor class of compounds. In the case of ondansetron, these effects have been rare and transient and noted primarily with IV administration, however, the extent to which ondansetron prolongs the QT interval has not been defined.

This study will quantify the effects of a single dose of IV ondansetron administered over 15 minutes on cardiac conduction in a double-blind, cross-over study and compared to placebo and a positive control, oral moxifloxacin. Pre- and post-dose digital electrocardiograms (ECGs) will be obtained by continuous Holter monitoring (1000 Hz) for blinded over-read by a third party vendor. This double-blind study will randomize approximately 60 healthy adult male and female volunteers to one of 12 sequences each consisting of 4 study treatment periods in a crossover design with a 7-day washout between each treatment period. Subjects will receive placebo, moxifloxacin (single 400 mg tablet), ondansetron 8 mg, and ondansetron 32 mg based on the randomized sequence. Both ondansetron and the placebo for ondansetron will be administered intravenously over 15 minutes. Moxifloxacin, a drug known to cause mild QTc prolongation, is included as a positive control and will be dosed as open label. Serial blood samples will be obtained to determine ondansetron and, if needed, moxifloxacin pharmacokinetic parameters. Safety and tolerability will be assessed through physical exams, adverse events, concurrent medications, clinical laboratory tests and vital signs.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult men and women, non-smokers between 18 and 45 years of age inclusive, at the time of signing the informed consent. Every effort will be made to enrol an approximately equal number of males and females.
* Signed and dated written informed consent prior to admission to the study, which includes compliance with the requirements and restrictions listed in the consent form.
* Healthy as judged by a responsible physician, with no clinically significant abnormality identified on the medical or laboratory evaluation performed at Screening, including 12-lead ECG. A subject with a clinical abnormality or laboratory parameters outside the reference range for this age group may be included only with the approval of the GSK medical monitor.
* ALT, alkaline phosphatase and bilirubin less than or equal to 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* A female is eligible to enter and participate in this study if she is of: Non-childbearing potential (i.e., physiologically incapable of becoming pregnant), including any female who either has had a hysterectomy or has had a bilateral oophorectomy (ovariectomy) or is post-menopausal defined as being amenorrhoeic for greater than or equal to 1 year with an appropriate clinical profile, e.g., age appropriate, history of vasomotor symptoms. Follicle-stimulating hormone (FSH) must be greater than or equal to 40 mIU/mL to confirm the post-menopausal state.

If a female is of child-bearing potential, has a negative serum pregnancy test at Screening, and agrees to or has undergone one of the following: Complete abstinence from sexual intercourse from 2 weeks prior to administration of the study drug until completion of the follow-up procedures, or, bilateral tubal ligation, or have a vasectomized partner or use an intrauterine device with published data showing that expected failure rate is less than 1% per year (e.g., GynaeFix) from 2 weeks prior to administration of study drug until completion of the follow-up procedures, or, use double-barrier method [condom or occlusive cap (diaphragm or cervical/vault caps) used with spermicidal foam/gel/cream/suppository].

* Body Mass Index (BMI)* in the range of 19 - 30 kg/m2 (inclusive). *[BMI = weight [kg]/(height [m])2]

Exclusion Criteria:

* Cardiac conduction abnormalities denoted by any of the following at screening:

QTc interval > 450 msec; PR interval > 240 msec or less than or equal to 110 msec; evidence of second- or third-degree atrioventricular (AV) block; pathological Q-waves (defined as Q-wave > 40 msec or depth greater than 0.4 - 0.5 mV); evidence of ventricular pre-excitation; electrocardiographic evidence of complete left bundle branch block, right bundle branch block (RBBB), incomplete LBBB; intraventricular conduction delay with QRS duration > 120 msec; bradycardia as defined by sinus rate < 50 bpm.

* Any history of myocardial infarction, syncope, long-QT syndrome, cardiac arrhythmias, or a history of uncontrolled hypertension or unstable heart disease within the 6 months prior to the screening visit, or a family history of long-QT syndrome or a family history of sudden death.
* Family history of heart attack or stroke at age less than or equal to 60 years.
* Levels of potassium, magnesium, and calcium outside the normal reference range at screening.
* Clinically significant serum chemistry and complete blood count parameters outside the normal reference range at screening.
* Positive for HIV antibody, hepatitis B virus S-antigen (HbSAg) or hepatitis C (Hep C) virus antibody at screening.
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* History of alcohol/drug abuse or dependence within 12 months of the study.
* History of regular alcohol consumption within 6 months of the study defined as: an average weekly intake of >14 drinks for males or >7 drinks for females. One drink is equivalent to 12 g of alcohol: 12 ounces (360 mL) of beer, 5 ounces (150 mL) of wine or 1.5 ounces (45 mL) of 80 proof distilled spirits.
* A positive pre-study urine test for drugs of abuse including alcohol at screening or prior to the start of dosing. A minimum list of drugs that will be screened for includes amphetamines, barbiturates, cocaine, opiates, cannabinoids, benzodiazepines, and cotinine. Subjects will be re-screened at each treatment period.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than 4 new chemical entities within 12 months prior to the first dosing day.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK medical monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* The subject has donated blood or blood products in excess of 500 mL within a 56 day period.
* Pregnant females as determined by positive serum hCG test at screening.
* Consumption of aspirin, aspirin-containing compounds, salicylates or nonsteroidal anti-inflammatory agents (NSAIDs) within 14 days of the study start and until the end of the follow-up visit. Acetaminophen (less than or equal to 2 g/day) will be permitted during the study for analgesia.
* Subject has consumed liquid antacids (e.g., Maalox, Mylanta, Amphojel, Milk of Magnesia) or chewable antacids (e.g., TUMS™) within 48 hours of the first dose of study medication, and throughout the duration of study drug administration.
* History of sensitivity to moxifloxacin or any member of the quinolone class of antimicrobial agents, or history of drug or other allergy that, in the opinion of the physician responsible, contraindicates their participation. If use of an IV cannula with heparinized flush is anticipated for PK draws, then hypersensitivity to heparin is also exclusionary.
* Urinary cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
* Consumption of red wine, seville oranges, grapefruit or grapefruit juice, pomelos, exotic citrus fruits, grapefruit hybrids or fruit juices from 7 days prior to the first dose of study medication.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2011-08-16 (Actual); Primary Completion 2011-12-19 (Actual); Study Completion 2011-12-19 (Actual)

PRIMARY OUTCOMES:
Change in QTcF after a single dose of Ondansetron given IV over 15 minutes. | Single dosing day at each of the 4 treatment periods with a 7-day washout between each period. The total duration of each subject's participation in the study, from screening through follow-up will be an average of 11 weeks.
  Two doses of ondansetron willl be used, 8mg and 32mg. The change in QTcF will be time-matched, baseline adjusted and compared to placebo.

SECONDARY OUTCOMES:
characterize relationship between changes in ddQTc and plasma concentrations of ondansetron | Single dosing day at each of the 4 treatment periods with a 7-day washout between each period. The total duration of each subject's participation in the study, from screening through follow-up will be an average of 11 weeks.
  The slope of the relationship between ddQTc and plasma ondansetron concentrations and predicted change in ddQtc will be used to determine.
characterize relationship between QT interval and plasma ondansetron | Single dosing day at each of the 4 treatment periods with a 7-day washout between each period. The total duration of each subject's participation in the study, from screening through follow-up will be an average of 11 weeks.
  The slope of the relationship between QTc interval and ondansetron concentrations and predicted change in QTc from baseline will be used to determine.
characterize the effect on QTcI and QTcB relative to placebo between the two doses of ondansetron and moxifloxacin | Single dosing day at each of the 4 treatment periods with a 7-day washout between each period. The total duration of each subject's participation in the study, from screening through follow-up will be an average of 11 weeks.
  ECG parameters will be measured and used to calculate this effect.
characterize effect on QT and HR relative to placebo of the two doses of ondansetron and moxifloxacin. | Single dosing day at each of the 4 treatment periods with a 7-day washout between each period. The total duration of each subject's participation in the study, from screening through follow-up will be an average of 11 weeks.
  ECG parameters will be measured along with vitals and used to calculate this effect.
characterize the pharmacokinetics of ondansetron. | Single dosing day at each of the 4 treatment periods with a 7-day washout between each period. The total duration of each subject's participation in the study, from screening through follow-up will be an average of 11 weeks.
  plasma concentrations of ondansetron will be measured and PK parameters (AUC, Cmax, tmax) determined.
characterize safety and tolerability of the two doses of ondansetron. | Single dosing day at each of the 4 treatment periods with a 7-day washout between each period. The total duration of each subject's participation in the study, from screening through follow-up will be an average of 11 weeks.
  Tolerability and safety will be assessed by 12-lead ECGs, telemetry, BP, HR, Adverse Events and clinical laboratory tests.
characterize the pharmacokinetics of moxifloxacin if needed. | Single dosing day at each of the 4 treatment periods with a 7-day washout between each period. The total duration of each subject's participation in the study, from screening through follow-up will be an average of 11 weeks.
  plasma concentrations of moxifloxacin will be measured and PK parameters (AUC, Cmax, tmax) determined if needed.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Austin, Texas, United States

REFERENCES:
- See also: Results for study 115458 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/115458?search=study&study_ids=115458#rs